CLINICAL TRIAL: NCT05568576
Title: Metabolic Syndrome and Long-term Survival Following Liver Resection for Hepatocellular Carcinoma Among Patients With Chronic Hepatitis C Virus Infection
Brief Title: Metabolic Syndrome and Long-term Survival Following Liver Resection
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Abu Elfatth, Lecturer of Tropical Medicine and Gastroenterology, Assiut University
Other Study IDs: ahmedtoH3
Record Dates: First submitted 2022-10-02; First posted 2022-10-05 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Survival
Keywords: Metabolic syndrome, survival, hepatocellular carcinom
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- patients with HCC underwent resection: patients with HCC underwent resection

SUMMARY:
Although hepatitis C virus (HCV) infection remains one of the main causes of hepatocellular carcinoma (HCC) worldwide, metabolic syndrome, with its increase in prevalence, has become an important and significant risk factor for HCC

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) represents the sixth most common cancer worldwide. In Egypt, it represents the fourth common cancer. Many hospital-based studies reported increasing the incidence of HCC. The reason for increased incidence could be attributed to (1) improvement in screening programs and diagnostic tools, (2) increasing the survival rate of cirrhotic patients that increases the chance of developing HCC, and (3) increasing the incidence and complications of hepatitis C virus (HCV) which is the most important risk factor in developing liver cancer including HCC in Egypt Precise staging of HCC initially is very useful for determination of the therapeutic options and the overall prognosis of the disease. There are certain clinical features upon which most staging systems use for HCC assessment. These clinical features are size and local extent of the tumor, metastasis of the tumor, severity of the liver disease, and the overall patient performance status Several studies in the United States, Europe, Taiwan, Hong Kong , and New Zealand have examined the potential relationships between various metabolic factors and HCC risks, mostly focusing on type 2 DM and obesity. Diabetes , or even prediabetes, has been observed to be a major metabolic factor related to an increased risk of HCC in individuals with HBV infections.

There is paucity in literature about effect of metabolic syndrome on Long-term Survival Following Liver Resection for Hepatocellular Carcinoma Among Patients With Chronic Hepatitis C Virus Infection

ELIGIBILITY:
Inclusion Criteria:

- All patients with HCC secondary to HCV infection underwent hepatic resection

Exclusion Criteria:

HBV patients other modalities of therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with HCC secondary to HCV infection underwent hepatic resection
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Survival | between two and five years
  assess frequency long term survival after resection

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Shwakt, Study Chair — Assiut University
Locations (1):
- Ahmed Mohammed Abu-Elfatth, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
with special request

REFERENCES:
- [Result] Tan Y, Zhang X, Zhang W, Tang L, Yang H, Yan K, Jiang L, Yang J, Li C, Yang J, Wen T, Tang H, Yan L. The Influence of Metabolic Syndrome on the Risk of Hepatocellular Carcinoma in Patients with Chronic Hepatitis B Infection in Mainland China. Cancer Epidemiol Biomarkers Prev. 2019 Dec;28(12):2038-2046. doi: 10.1158/1055-9965.EPI-19-0303. Epub 2019 Sep 18. PMID 31533942
- [Result] Rashed WM, Kandeil MAM, Mahmoud MO, Ezzat S. Hepatocellular Carcinoma (HCC) in Egypt: A comprehensive overview. J Egypt Natl Canc Inst. 2020 Jan 16;32(1):5. doi: 10.1186/s43046-020-0016-x. PMID 32372179